CLINICAL TRIAL: NCT03067506
Title: A Single Center Pilot Study to Evaluate Real Time Passive and Active High-Frequency Cognitive and Mood Assessment Data in Major Depressive Disorder Using Digital Wearable Technology
Brief Title: Cognitive and Mood Assessment Data in Major Depressive Disorder Using Digital Wearable Technology
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: MDD-5003
Record Dates: First submitted 2017-02-26; First posted 2017-03-01 (Actual); Results first posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-07

CONDITIONS: Major Depressive Disorder
Keywords: Drug Therapy
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With Major Depressive Disorder (MDD): Participants with MDD were provided with an Apple watch on which brief cognitive and mood tests were evaluated daily up to 6 weeks.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study was to evaluate the feasibility and compliance with a novel method for assessing mood and cognition in participants with major depressive disorder (MDD).

DETAILED DESCRIPTION:
The novel method being tested in this study for assessing mood and cognition in participants with MDD was wearable technology. This study looked at the correlation of mood and cognition outcomes on wearable technology with traditional objective neuropsychological cognitive function tests and self-reported mood outcomes.

The study enrolled approximately 30 patients. Participants were provided with a watch on which brief cognitive and mood tests were evaluated daily up to 6 weeks.

All participants prompted to complete cognitive and mood assessments on 3 occasions across the day. Two occasions (morning and afternoon) comprised assessment of cognition, and the final assessment in the evening constituted a review of the day focusing on self-reported depressed mood.

This single-center trial was conducted in United Kingdom. The overall time to participate in this study was 6 weeks. Participants took part up to 5 study visits (1 in-person on-site visit, 3 web-based and 1 at home visit) assessing performance on traditional objective neuropsychological cognitive function tests and self-reported measures of depression symptom severity and social function.

ELIGIBILITY:
Inclusion Criteria:

1. Has MDD as the primary psychiatric diagnosis.
2. Has been treated previously with at least 1 antidepressant (monotherapy).
3. Has scores on Participant Health Questionnaire-9 items (PHQ-9) ≥5 and PHQ-9 ≤15 at Screening

Exclusion Criteria:

1. Has a significant risk of suicide according to the investigator's clinical judgment or has made an actual suicide attempt in the previous 6 months prior to Screening.
2. Has a history of only responding to either combination or augmentation therapy in the current episode and has had been treated for more than a year without any period of remission.
3. Has 1 or more of the following:

   1. Current or history of: manic or hypomanic episode, schizophrenia or any other psychotic disorder, including schizoaffective disorder, major depression with psychotic features, bipolar depression with psychotic features, obsessive compulsive disorder, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5).
   2. Current diagnosis or history of alcohol or other substance abuse or dependence (excluding nicotine or caffeine).
   3. Neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with major depressive disorder (MDD) were provided with an Apple watch on which brief cognitive and mood tests were evaluated daily up to 6 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Takeda Investigative Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United Kingdom from 29 February 2017 to 03 July 2017.
Pre-assignment Details: Participants with a diagnosis of major depressive disorder (MDD) prescribed first-, second- or third-line antidepressant monotherapy were provided with an Apple watch on which brief cognitive and mood tests were evaluated.
Period: Overall Study
Arm/Group | Participants With Major Depressive Disorder (MDD)
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants with major depressive disorder (MDD) who were enrolled in the study.
Arm/Group | Participants With Major Depressive Disorder (MDD)
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.23 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 30
Screening Patient Health Questionnaire-9 items (PHQ 9) [Mean (Standard Deviation); unit: score on a scale] — PHQ-9 is a 9-items scale to assess depression. Each item is rated (0=not at all to 3=nearly every day) for total score 0-27 (higher scores indicate severe depression).
  score on a scale | 9.13 (3.13)
Comorbid Anxiety [Number; unit: participants] | 20
Current Medication [Number; unit: participants]
  Amitriptyline | 4
  Citalopram | 9
  Escitalopram | 1
  Fluoxetine | 2
  Mirtazapine | 2
  Sertraline | 8
  Trazodone | 1
  Venlafaxine | 3
Current Medication by Category [Number; unit: participants]
  Serotonin Antagonist and Reuptake Inhibitor (SARI) | 1
  Serotonin-Norepinephrine Reuptake Inhibitor (SNRI) | 5
  Selective Serotonin Reuptake Inhibitor (SSRI) | 20
  Tricyclic Antidepressant (TCA) | 4
Time on Current Medication [Mean (Standard Deviation); unit: months] | 9.93 (9.74)
Medical Switch [Number; unit: participants] | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days on Which Daily N-back Sessions Were Completed
Description: The cognitive assessment n-back test was completed on the wearable technology (Apple watch) on 3 occasions across the day in the morning, afternoon and evening.
Time Frame: Baseline up to Week 6
Population: Analysis population included all participants with major depressive disorder (MDD) who were enrolled in the study.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Participants With Major Depressive Disorder (MDD)
Number analyzed (Participants) | 30
percentage of days | 95.63 (9.28)

2. Primary Outcome: Percentage of Days on Which Daily Mood Assessment Tests Were Completed
Description: The Daily Mood assessments were completed on the wearable technology (Apple watch) once per day in the afternoon or evening.
Time Frame: Baseline up to Week 6
Population: Analysis population included all participants with major depressive disorder (MDD) who were enrolled in the study.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Participants With Major Depressive Disorder (MDD)
Number analyzed (Participants) | 30
percentage of days | 94.6 (9.73)

3. Primary Outcome: Correlation Coefficient Between Measures of Cognition (N-back Scores) and Performance on the Cambridge Neuropsychological Test Automated Battery (CANTAB) Tests: Spatial Working Memory Between Errors (SWMBE) and Spatial Working Memory Strategy (SWMS)
Description: The n-back was used to assess cognition 3 times a day. Participants responded by touching the watch face when a symbol matched the one presented 2-back. Average daily n-back score (d-prime) was calculated.
  CANTAB tests consists of a battery of neuropsychological tests. Spatial Working Memory (SWM) assessed retention of spatial data, ability to manipulate remembered items and strategize. Participant was asked to find tokens in on-screen boxes and move them.
  SWMBE=cumulative number of times participant went back to box that a token was previously removed per each successful study. Lower score was better.
  SWMS=number of unique boxes participant searched in two 6 and 8 box trials. Total of 4 trial scores ranged from 4-28. Lower score indicated better performance.
  Pearson's correlation coefficient measured linear correlation between n-back scores from Apple Watch and CANTAB tests, provided as a value +1=positive correlation to -1=negative correlation. 0=no correlation.
Time Frame: Baseline up to Week 6
Population: Analysis population included all participants with major depressive disorder (MDD) who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: Correlation Coefficient (r)
Arm/Group | Participants With Major Depressive Disorder (MDD)
Number analyzed (Participants) | 30
Correlation Coefficient (r)
  SWMBE | -0.46 [-0.70 to -0.11]
  SWMS | -0.37 [-0.65 to -0.01]

4. Primary Outcome: Correlation Coefficient Between Measures of Cognition (N-back Scores) and Performance on the CANTAB Test: Rapid Visual Information Processing (RVP)
Description: The n-back was used to assess cognition 3 times a day. Participants responded by touching the watch face when a symbol matched the one presented 2-back. Average daily n-back score (d-prime) was calculated.
  CANTAB tests consists of a battery of neuropsychological tests. RVP measures sustained attention. A white box appears in the center of the computer screen, inside which digits, from 2 to 9, appear in a pseudo-random order, at the rate of 100 digits per minute. Participants are requested to detect target sequences of digits.
  RVPA=measure of sensitivity to the target, regardless of response tendency (expected range is 0.00 to 1.00).
  Speed of Processing (RVPMDL)=The mean response latency during assessment sequence blocks where the participant responded correctly.
  Pearson's correlation coefficient measured linear correlation between n-back scores from Apple Watch and CANTAB tests, provided a value +1=positive correlation to -1=negative correlation. 0=no correlation.
Time Frame: Baseline up to Week 6
Population: Analysis population included all participants with major depressive disorder (MDD) who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: Correlation Coefficient (r)
Arm/Group | Participants With Major Depressive Disorder (MDD)
Number analyzed (Participants) | 30
Correlation Coefficient (r)
  RVPA (Sensitivity to Target) | 0.50 [0.17 to 0.73]
  RVPMDL (Speed of Processing) | -0.40 [-0.67 to -0.04]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 6
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Participants With Major Depressive Disorder (MDD)
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT03067506/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT03067506/SAP_001.pdf